CLINICAL TRIAL: NCT03296748
Title: Is There Any Value of Concomitant Repair of Asymptomatic Grade II Anterior Vaginal Wall Prolapse During Mid Urethral Sling Surgery for Stress Urinary Incontinence ?
Brief Title: Correction of Asymptomatic 2nd Degree Cystocele in Patient With Stress Incontinence
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, sarah mohamed hassan, lecturer of obstetrics and gynecology Cairo university, Kasr El Aini Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 151115
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Stress Urinary Incontinence
Keywords: asymptomatic cystocele.; stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: female patients with stress urinary incontinence and asymptomatic grade II anterior vaginal wall prolapse were divided into Group A: treated only with trans-obturator tape (TOT) and group B where' TOT was associated with anterior colporrhaphy .
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TOT only group (Active Comparator): 60 patients with stress incontinence and asymptomatic grade 2 cystocele.
  Interventions: Procedure: trans-obturator tape inside-out usingsoft tapes.
- concomitant repair group (Active Comparator): 63 patients with stress incontinence and asymptomatic grade 2 cystocele.
  Interventions: Procedure: trans-obturator tape inside-out usingsoft tapes.; Procedure: anterior colporraphy

INTERVENTIONS:
Procedure: trans-obturator tape inside-out usingsoft tapes. — trans-obturator tape inside-out soft tapes is applied under spinal anesthesia. After the procedure, the vaginal gauze packing and Foley catheter were removed on the morning of the next day.
  Other Names: anterior colporrhaphy
Procedure: anterior colporraphy
  Arms: concomitant repair group

SUMMARY:
The aim of our study is to assess the value of concomitant surgical correction of asymptomatic grade II anterior vaginal wall prolapse with the placement of midurethral sling for treatment of female patients with stress incontinence

DETAILED DESCRIPTION:
female patients with stress urinary incontinence and asymptomatic grade II anterior vaginal wall prolapse were divided into Group A: treated only with trans-obturator tape (TOT) and group B where' TOT was associated with anterior colporrhaphy and the outcome is compared.

ELIGIBILITY:
Inclusion Criteria:

* female patients
* genuine stress incontinence

  * asymptomatic cystocele

Exclusion Criteria:

* mixed incontinence

Ages: 23 Years to 56 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
cure rate of stress incontinence | 3 months after surgery
  by clinical assessment
Denovo urgency | 3 months after surgery
  by clinical assessment

SECONDARY OUTCOMES:
cure rate of stress incontinence | 6 months after surgery
  by clinical assessment
cure rate of stress incontinence | 12 months after surgery
  by clinical assessment
Denovo urgency | 6 months after surgery
  by clinical assessment
Denovo urgency | 12 months after surgery
  by clinical assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainiy Hospital, Cairo, Egypt